CLINICAL TRIAL: NCT06995170
Title: Investigation of the Correlation Between Polyamine Levels and Their Key Enzymatic Activities in Association With Inflammatory Bowel Disease Progression
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20242438
Record Dates: First submitted 2025-04-14; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease; Polyamines; Infliximab
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — fecal ,plasma, urine and fixed tissue samples of some participants will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- IBD group: IBD patients aged 18-65 years were categorized into remission and active-phase groups according to corresponding clinical scoring scales. IBD patients will be recruited from The First Affiliated Hospital of the Air Forth Medical University from January 2025 to December 2025.
- Healthy subjects: Age-, gender-, and education level-matched healthy controls will be recruited from The First Affiliated Hospital of the Air Forth Medical University from January 2025 to December 2025.
- First-line biologics group: 18-65-year-old Inflammatory Bowel Disease (IBD) patients planned for the first administration of Infliximab will be recruited from The First Affiliated Hospital of the Air Forth Medical University from January 2025 to December 2025.

SUMMARY:
Inflammatory Bowel Disease (IBD), encompassing Ulcerative Colitis (UC) and Crohn's Disease (CD), significantly impairs patients' quality of life. Current monitoring of disease activity primarily relies on endoscopy combined with histological examination, which is associated with high costs, invasiveness, poor patient tolerance, and risks of complications. Additionally, disease activity indices and laboratory-based IBD staging metrics demonstrate limited utility and accuracy in clinical practice. This study aims to investigate the correlation between polyamine levels and their key enzymes in the polyamine metabolism pathway with IBD activity, thereby establishing a predictive model for IBD progression through polyamine and metabolite measurements; to estimate the efficacy of biologics via polyamine detection, providing a scientific basis for therapeutic selection; and to screen gut microbiota associated with polyamine metabolic alterations, offering evidence-based guidance for probiotic selection in IBD patients.

DETAILED DESCRIPTION:
According to the inclusion and exclusion criteria, 91 patients with IBD diagnosed in the Department of Gastroenterology, the First Affiliated Hospital of Air Force Medical University from November 2024 to September 2025 were included, and the subjects were divided into remission group and active group according to the corresponding IBD scale scores; 46 healthy controls were generally included according to the number of patients; In addition, 47 patients in the first biologic treatment group were included according to the inclusion and exclusion criteria. The FFQ scale was used to calculate and evaluate the intake of polyamines in the enrolled patients, high performance liquid chromatography and mass spectrometry were used to measure the levels of polyamines in serum and fecal samples of patients, and immunohistochemical semi quantitative analysis of colon pathological sections was used to analyze the levels of key enzymes of polyamine metabolism.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years;
2. Diagnosed with inflammatory (IBD) according to the Chinese Guidelines for the Diagnosis and Treatment of Ulcerative Colitis (2023, Xi'an) and the Chinese Guidelines for the Diagnosis and Treatment of Crohn's Disease (2023, Guangzhou);
3. Complete medical records available and written informed consent obtained from the participant.

Exclusion Criteria:

1. Presence of other metabolic disorders;
2. History of malignant tumors, severe organ dysfunction, or other severe systemic diseases affecting major organs, or hematological disorders;
3. Diagnosis of influenza, bacterial dysentery, or other infectious diseases within the past 2 weeks;
4. Presence of other diseases that may interfere with polyamine metabolism;
5. Use of antibiotics or probiotics within 8 weeks prior to the start of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IBD patients aged 18-65 years were recruited from The First Affiliated Hospital of the Air Forth Medical University.
Sampling Method: Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disease activity | at baseline
  For patients with recent colonoscopy results: UC patients are assessed for disease activity using the modified Mayo score, while CD patients are evaluated using the SECA score.
  For patients without recent colonoscopy results: UC patients are assessed for disease activity using the Modified Truelove and Witts Grading System, and CD patients are evaluated using the SCAI for disease activity assessment.
  The modified Mayo score:Clinical remission is defined as a total score of ≤2 points and no single sub-item score >1. Mild activity is defined as 3-5 points, moderate activity as 6-10 points, and severe activity as 11-12 points.
  SECA:0 ~ 2 Indicates endoscopic remission,3 ~ 6 suggests mild disease activity,7 ~ 15 indicates moderate disease activity,≥16 reflects severe disease activity.
  SCAI: Total score ≤4: Indicates endoscopic remission. 5-7: Suggests mild disease activity. 8-16: Reflects moderate disease activity. >16: Signifies severe disease activity.
The level of polyamine | at baseline and 8weeks
  The levels of putrescine, spermidine, N1-acetylspermidine, ornithine, citrulline, N1-acetylspermidine, N1-acetylspermine, N8-acetylspermidine, N-acetylornithine, N1,N12-diacetylspermine, and N-acetylputrescine in serum, feces, and urine are measured using mass spectrometry. Results will be reported in nmol/L, with levels potentially reflecting disease activity.
Food Frequency Questionnaire | at baseline
  Including 9 food groups and 59 food items. The patient's total monthly polyamine intake is calculated by multiplying the total monthly consumption of each food item by its corresponding polyamine content.Total polyamine intake (mg/month) = Σ (Food consumption [g/month] × Polyamine content [mg/g])
Gastrointestinal Microbiome | at baseline
  Fecal samples of some participants will be collected and prepared. DNA will be extracted from the stool samples, and the V3-V4 hypervariable region of bacterial 16S rRNA gene was sequenced.

SECONDARY OUTCOMES:
polyamine metabolic enzymes | at baseline
  Intestinal mucosal sections were stained with immunohistochemistry to quantify the content and distribution of the key polyamine metabolic enzyme Ornithine Decarboxylase (ODC).

CONTACTS AND LOCATIONS:
Overall Officials: Kaichun Wu, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No